CLINICAL TRIAL: NCT00373412
Title: Randomized, Phase 1 Trial to Evaluate Safety and CMV-Specific Immune Response to a pDNA CMV Trivalent Vaccine (VCL-CT02) Followed by Towne CMV Vaccine (Towne) Challenge in Healthy, CMV- Seronegative Adults
Brief Title: Trial of pDNA CMV Vaccine (VCL-CT02) Followed by Towne CMV Vaccine (Towne) Challenge
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Vical (Industry)
Responsible Party: Mark Jacobson, Professor of Medicine, UCSF
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Jacobson VCL CT-02 TC
Record Dates: First submitted 2006-09-06; First posted 2006-09-08 (Estimated); Last update posted 2008-05-08 (Estimated); Status verified 2006-10

CONDITIONS: Cytomegalovirus Infection
Keywords: cytomegalovirus; vaccine; T cell; antibodies
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: VCL CT02 pDNA vaccine
Biological: Towne CMV vaccine

SUMMARY:
Objectives of this trial are to:

Evaluate the kinetics and magnitude of the CMV-specific immune response post-Towne challenge (3000 pfu) in healthy CMV-seronegative volunteers who receive VCL CT02 administered (1 mg weekly x 3) 3 months previously compared to randomized controls who do not receive VCL CT02 as measured by:

1. antibody titers for gB;
2. T-cell IFN-g ELISPOT;
3. T-cell proliferation assays for IE1, pp65, and/or gB; and
4. cytokine and phenotypic flow cytometry responses to pp65, IE1, and/or gB.

Evaluate the safety safety of Towne challenge in healthy CMV-seronegative adult subjects who have previously been immunized with a trivalent pDNA CMV vaccine (VCL-CT02) administered intramuscularly.

Our hypothesis is that the immune response to Towne vaccine 3000 pfu challenge after VLC-CT02 priming will be greater than that after Towne vaccination alone.

DETAILED DESCRIPTION:
This is a Phase 1, single-center, randomized, open-label trial of the live, attenuated Towne CMV vaccine administered as a "challenge" to healthy, CMV-seronegative, adult subjects who previously receive the CMV immunotherapeutic trivalent pDNA-based vaccine, VCL-CT02, given by intramuscular route at Days 1, 7 and 14 or who receive no VCL-CT02.

Up to 12 healthy, CMV-seronegative subjects will be enrolled. If a subject consents and meets all eligibility criteria, the subject will be randomized to the VCL CT02 (N=6)or control (N=6) groups. VCL CT02-assigned subjects will receive VCL CT02 (1 mg weekly x 3) and then on Day 77 will received Towne vacine (3000 pfu subcutaneously). Control-assigned subjects will receive Towne alone. Safety will be monitored and both antibody to CMV gB and T-cell responses to CMV antigens will be measured at specified intervals for 252 days post Towne challenge.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 45 years of age
* Normal lab values at study entry
* Good general health
* Negative CMV IgG antibody test

Exclusion Criteria:

* CMV seropositive
* Recent vaccination(s)
* Immunodeficiency
* Vaccination with investigational CMV vaccine(s)
* Pregnant or breast-feeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16
Dates: Start 2006-10; Primary Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
CMV-specific immune response post-Towne challenge: gB antibody, T-cell IFN-g ELISPOT, T-cell proliferation assays for IE1, pp65, and/or gB, cytokine and phenotypic flow cytometry responses to pp65, IE1, gB.

SECONDARY OUTCOMES:
Safety of Towne challenge in subjects who have previously been immunized with a trivalent pDNA CMV vaccine (VCL-CT02).

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Jacobson, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Positive Health Program, 995 Potrero, 4th Floor, San Francisco, California, United States